CLINICAL TRIAL: NCT06514599
Title: Comparison of The Efficacy of CRP, Procalcitonin and Pro-BNP as Diagnostic and Prognostic Markers in AECOPD
Brief Title: CRP, Procalcitonin and Pro-BNP as Diagnostic and Prognostic Markers in AECOPD
Acronym: AECOPD
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Serkan Doğan, Assoc. Prof., Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2023.02.21
Record Dates: First submitted 2024-07-10; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: COPD Exacerbation Acute
Keywords: COPD; pro-BNP; procalcitonin; exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD) are one of the chief causes for admission to Emergency Department. AECOPD is a significant cause for mortality and morbidity worldwide. Emergency Medicine Physicians frequently manage these patients. Predicting the severity and possible prognosis of AECOPD is an important task for Emergency Medicine Physicians as treatment options and aggressiveness may depend on these predictions. In our study we aimed to compare different biomarkers such as Procalcitonin, Pro-Brain Natriuretic Peptide (Pro-BNP) and C-Reactive Protein (CRP) on their efficacy at predicting the severity and prognosis of AECOPD.

We analyzed the data of the selected 196 patients with the diagnosis AECOPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2024 guide who were admitted to our Emergency Department between 15/02/2023 and 15/02/2024.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is an important health concern worldwide and causes serious mortality and morbidities. Although prevalences can differ across different countries, it was predicted that 480 million people are affected from COPD in 2020 alone (1).

COPD is a condition that is characterized by an irreversible chronic inflammation which occurs within the airways, the pulmonary vasculature and parenchyma of the lungs. As a part of the progress of this disease, cough, dyspnea and sputum production could become almost permanent as symptoms. Furthermore, depending on seasonal changes, COPD can present itself with exacerbations, lowering the life quality of the patient and potentially overloading the healthcare systems across the world.

COPD exacerbations influence the general condition of the patient. They can cause admittance rates of COPD patient to significantly increase. They can also cause mortalities as well. A COPD patient can have a 5-year mortality rate of up to %50 if they are hospitalized with a COPD exacerbation (2). COPD exacerbations are diagnosed with a detailed medical history, physical examination and necessary diagnostic tests. According the GOLD 2024 guidelines, in order to diagnose and classify a patient with a preliminary diagnosis of a COPD exacerbation Visual Analogue Scale (VAS) dyspnea score, respiratory rate, heart rate, resting oxygen saturation, arterial blood gas and C-reactive protein (CRP) levels are among these necessary diagnostic tests.

There are studies mentioning CRP and Procalcitonin levels as independent diagnostic biomarkers for asthma and COPD exacerbations (3). There are also studies with findings that support the idea of using CRP and Procalcitonin levels as independent biomarkers to guide the antibiotic therapy in these patients (3-6). In addition to these markers, Pro Brain Natriuretic Peptide (Pro-BNP) is found to be a potentially effective biomarker in predicting the prognosis of COPD patients, both independently and alongside other cardiac biomarkers in a number of studies (7).

In this study we have aimed to compare the efficacy of CRP, Procalcitonin and Pro-BNP as diagnostic and prognostic markers in COPD patients. We focused specifically on Procalcitonin and Pro-BNP and if there is any potential superiority of these biomarkers against CRP while evaluating COPD exacerbation patients.

This prospective and observational study was conducted in an emergency department (ED) of a tertiary care referral center for the western part of Istanbul. Approximately 80-100 patients with various types of life-threatening emergencies daily receive healthcare service in the red area of the ED. Respiratory distress, dyspnea, and acute lung diseases are leading causes of emergency admission in our department. Our ED involved fully equipped and well-qualified critical care unit and resuscitation areas to provide urgent care and life-saving interventions for those patients. Thus, this study was conducted under optimal infrastructural conditions for patients with COPD exacerbation.

The patients for this study were recruited in the ED between 15/02/2023-15/02/2024. In order to form a database to use for our research, a data collection form was organized for each individual. This form compromised of the patient's saturation without supplemental oxygen, heart rate in beats per minute, blood pressure with both systolic and diastolic values separately recorded, body temperature, Electrocardiogram and respiratory rate, with all of them being measured at admittance. A detailed medical history, including the previous and chronic diseases, prescription medicines, past surgeries or invasive procedures and smoking habits, were also added to this data collection form.

ELIGIBILITY:
Inclusion Criteria:

* being older than 18 years old
* having been diagnosed with COPD by a specialist
* fulfilling the definition of an exacerbation set by GOLD 2024 guide which are having increased dyspnea, cough and sputum in a timespan of less than 14 days with or without tachypnea and tachycardia
* having signed the consent and approval form.

Exclusion Criteria:

* being younger than 18 years old
* not having been diagnosed with COPD by a specialist, not fulfilling the definition of an exacerbation set by GOLD 2024 guide
* refusing to sign the consent and approval form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients for this study were recruited in the ED between 15/02/2023-15/02/2024.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Attack Severity | At admission
  Mild, Moderate and Severe

SECONDARY OUTCOMES:
Mortality | 28 days
  AECOPD-related death

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, University of Health Sciences, İstanbul Kanuni SUltan Suleyman TRaining and Research Hospital, Istanbul, Küçükçekmece, Turkey (Türkiye)

REFERENCES:
- [Background] Boers E, Barrett M, Su JG, Benjafield AV, Sinha S, Kaye L, Zar HJ, Vuong V, Tellez D, Gondalia R, Rice MB, Nunez CM, Wedzicha JA, Malhotra A. Global Burden of Chronic Obstructive Pulmonary Disease Through 2050. JAMA Netw Open. 2023 Dec 1;6(12):e2346598. doi: 10.1001/jamanetworkopen.2023.46598. PMID 38060225
- [Background] Hoogendoorn M, Hoogenveen RT, Rutten-van Molken MP, Vestbo J, Feenstra TL. Case fatality of COPD exacerbations: a meta-analysis and statistical modelling approach. Eur Respir J. 2011 Mar;37(3):508-15. doi: 10.1183/09031936.00043710. Epub 2010 Jul 1. PMID 20595157
- [Background] Bafadhel M, Clark TW, Reid C, Medina MJ, Batham S, Barer MR, Nicholson KG, Brightling CE. Procalcitonin and C-reactive protein in hospitalized adult patients with community-acquired pneumonia or exacerbation of asthma or COPD. Chest. 2011 Jun;139(6):1410-1418. doi: 10.1378/chest.10-1747. Epub 2010 Oct 28. PMID 21030489
- [Background] Mathioudakis AG, Chatzimavridou-Grigoriadou V, Corlateanu A, Vestbo J. Procalcitonin to guide antibiotic administration in COPD exacerbations: a meta-analysis. Eur Respir Rev. 2017 Jan 31;26(143):160073. doi: 10.1183/16000617.0073-2016. Print 2017 Jan. PMID 28143877
- [Background] Colak A, Yilmaz C, Toprak B, Aktogu S. Procalcitonin and CRP as Biomarkers in Discrimination of Community-acquired Pneumonia and Exacerbation of COPD. J Med Biochem. 2017 Apr 22;36(2):122-126. doi: 10.1515/jomb-2017-0011. eCollection 2017 Apr. PMID 28680355
- [Background] Stolz D, Christ-Crain M, Bingisser R, Leuppi J, Miedinger D, Muller C, Huber P, Muller B, Tamm M. Antibiotic treatment of exacerbations of COPD: a randomized, controlled trial comparing procalcitonin-guidance with standard therapy. Chest. 2007 Jan;131(1):9-19. doi: 10.1378/chest.06-1500. PMID 17218551
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Wier LM, Elixhauser A, Pfuntner A, Au DH. Overview of Hospitalizations among Patients with COPD, 2008. 2011 Feb. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #106. Available from http://www.ncbi.nlm.nih.gov/books/NBK53969/ PMID 21510031
- [Background] Pantzaris ND, Spilioti DX, Psaromyalou A, Koniari I, Velissaris D. The Use of Serum Procalcitonin as a Diagnostic and Prognostic Biomarker in Chronic Obstructive Pulmonary Disease Exacerbations: A Literature Review Update. J Clin Med Res. 2018 Jul;10(7):545-551. doi: 10.14740/jocmr3458w. Epub 2018 Jun 4. PMID 29904438
- [Background] Zhu JJ, Liu LJ. Analysis of factors influenced by the effectiveness of non-invasive ventilation in the treatment of acute exacerbation of chronic obstructive pulmonary disease with different severities. Eur Rev Med Pharmacol Sci. 2016 Nov;20(22):4775-4781. PMID 27906423